CLINICAL TRIAL: NCT04418063
Title: Glenohumeral Internal Rotation Deficit in Non-pitcher Overhead Athletic Athletes: Case Series Analysis of Athletes
Acronym: GIRDAhtlFMUI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andri Maruli Tua Lubis, Principal Investigator, Indonesia University
Other Study IDs: GIRD-Ahtl-FMUI
Record Dates: First submitted 2020-05-31; First posted 2020-06-05 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Shoulder Injuries; Shoulder Syndrome; Injury;Sports; Sport Injury
Keywords: shoulder; glenohumeral internal rotation deficit; throwing athletic athlete
MeSH Terms: conditions — Shoulder Injuries; Athletic Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this observational case series the investigators would like to investigate wether or not the strenuous activity exerted on over head athletic athletes (ie. javelin throwers, discus throwers) may incite injury on their shoulders.

The investigators understood that these athletes had to perform repeated throwing motions and yet reports on their effects are very limited. This condition in the long run may contribute to injury and affecting performance of the athletes.

The investigators found that these relationships have not been looked at closely by others and largely overshadowed by athletes in other fields; such injury patterns had been described in details in baseball pitchers but not in other athletes.

DETAILED DESCRIPTION:
Description of protocol:

In this study, the investigators would recruit athletes from the national athletics federation training in our city.

Data collection:

History taking:

* complaints of shoulder stiffness
* need for prolonged warm-up
* pain
* discomfort relating to the shoulders

Physical examination:

* Bilateral shoulder range of motion (internal and external rotation)
* Posterior shoulder flexibility test (denotes internal rotation deficit)
* Scapular malpositioning, inferior medial border prominence, coracoid pain and malposition and dyskinesis of scapular movement (SICK) scapula rating

Notes: measurements are taken by at least two investigators separately and compared to ensure accuracy.

Results are presented in a table and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Performed overhead throwing motions in their athletic skills
* Athletes have competed in regional and national level
* Undergoing active training

Exclusion Criteria:

* Apparent anatomical deformity
* Sustaining injury(ies)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National athletic athletes that performed overhead throwing motion in their sports that meet the inclusion criteria within our city.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Glenohumeral internal rotation deficit | 1 day
  A deficit of >20 degrees between dominant and non-dominant shoulder

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol
Time Frame: The IPD will become available starting 6 months after publication.
Access Criteria: The information will be shared electronically via email to other researchers after review by the principal investigator.

REFERENCES:
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part I: pathoanatomy and biomechanics. Arthroscopy. 2003 Apr;19(4):404-20. doi: 10.1053/jars.2003.50128. PMID 12671624
- [Background] Burkhart SS, Morgan CD, Kibler WB. The disabled throwing shoulder: spectrum of pathology Part III: The SICK scapula, scapular dyskinesis, the kinetic chain, and rehabilitation. Arthroscopy. 2003 Jul-Aug;19(6):641-61. doi: 10.1016/s0749-8063(03)00389-x. No abstract available. PMID 12861203
- [Background] Keller RA, De Giacomo AF, Neumann JA, Limpisvasti O, Tibone JE. Glenohumeral Internal Rotation Deficit and Risk of Upper Extremity Injury in Overhead Athletes: A Meta-Analysis and Systematic Review. Sports Health. 2018 Mar/Apr;10(2):125-132. doi: 10.1177/1941738118756577. Epub 2018 Jan 30. PMID 29381423
- [Result] Rose MB, Noonan T. Glenohumeral internal rotation deficit in throwing athletes: current perspectives. Open Access J Sports Med. 2018 Mar 19;9:69-78. doi: 10.2147/OAJSM.S138975. eCollection 2018. PMID 29593438